CLINICAL TRIAL: NCT02248584
Title: SUPPLEMENTATION OF VITAMIN E, C and ZINC IN PATIENTS WITH NON-MELANOMA SKIN CANCER: INFLUENCE ON OXIDATIVE STRESS AND INFLAMMATORY STATE
Brief Title: VITAMIN E, C and ZINC IN PATIENTS WITH SKIN CANCER: INFLUENCE ON OXIDATIVE STRESS AND INFLAMMATORY STATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Responsible Party: Principal Investigator, Patricia Moriel, PhD, University of Campinas, Brazil
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Betania
Record Dates: First submitted 2014-09-22; First posted 2014-09-25 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Skin Neoplasms
MeSH Terms: conditions — Skin Neoplasms | interventions — Ascorbic Acid; Zinc

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Vitamin E, C and Zinc (Experimental): Capsule containing vitamin C (50 mg; CVS Quality, USA), vitamin E (60 mg; Nature´s Bounty, USA), and zinc (40 mg; CVS Quality, USA) per day for 60 days.
  Interventions: Dietary Supplement: Vitamin C, E and Zinc
- Placebo (Placebo Comparator): Capsule containing only lactose

INTERVENTIONS:
Dietary Supplement: Vitamin C, E and Zinc — Capsule containing vitamin C (50 mg; CVS Quality, USA), vitamin E (60 mg; Nature´s Bounty, USA), and zinc (40 mg; CVS Quality, USA) per day for 60 days.
  Arms: Vitamin E, C and Zinc

SUMMARY:
The objective of this study was to evaluate the effects of supplementary antioxidant therapy on the levels of biomarkers and inflamatory citocines in patients with a previous history of non-melanoma skin cancer treated with surgery. This was a double-blind, randomized, placebo-controlled trial. Patients were randomized into two groups, one receiving placebo (n=34) and the other receiving supplementary antioxidant therapy (n=26) with vitamin C (50 mg), vitamin E (60 mg), and zinc (40 mg) for 60 days. Blood samples were obtained from patients, and the levels of oxidative stress biomarkers, including 8-isoprostane, nitrite, thiobarbituric acid reactive substances, and total antioxidant capacity, were measured, as well as the inflamatory citocines (IL-1, IL-6, IL-10, TNF alfa) and it was evaluated at two different times: (1) one day before the start of supplementation or placebo administration and (2) at 60 days after intervention. Statistical analyses were performed with the SAS System for Windows 9.3 program and data were analyzed using ANOVA for repeated measures test.

ELIGIBILITY:
Inclusion Criteria:

* patients who had non-melanoma skin cancer (squamous cell carcinoma or basal cell carcinoma) and who were treated with surgery
* age ≥20 years
* absence of comorbidities such as type 1 diabetes, severe heart disease, hepatic dysfunction, renal failure requiring dialysis, HIV infection, and melanoma skin cancer
* no history of chemotherapy or radiotherapy in the previous 6 months
* absence of severe psychiatric disease that limited comprehension
* not taking any vitamin and/or mineral supplementation.

Exclusion Criteria:

* subjects did not complete the entire course of supplemental therapy.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
OXIDATIVE STRESS BIOMARKERS | one day before the start of supplementation or placebo administration and at 60 days after intervention
  8-isoprostane, Thiobarbituric Acid Reactive Substances (TBARS), Nitrite, Total Antioxidant Capacity (TAC)
INFLAMMATORY STATE | one day before the start of supplementation or placebo administration and at 60 days after intervention
  IL-1, IL-6, IL-10, TNF alfa

REFERENCES:
- [Derived] Freitas Bde J, Lloret GR, Visacri MB, Tuan BT, Amaral LS, Baldini D, de Sousa VM, de Castro LL, Aguiar JR, Pincinato Ede C, Mazzola PG, Moriel P. High 15-F2t-Isoprostane Levels in Patients with a Previous History of Nonmelanoma Skin Cancer: The Effects of Supplementary Antioxidant Therapy. Biomed Res Int. 2015;2015:963569. doi: 10.1155/2015/963569. Epub 2015 Oct 5. PMID 26509174